CLINICAL TRIAL: NCT01529970
Title: Genetic Study in Young Onset Parkinson's Disease
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: China Medical University Hospital (Other)
Responsible Party: Principal Investigator, Hui-Chun Huang, Attending Physician, China Medical University Hospital
Other Study IDs: DMR100-IRB-252
Record Dates: First submitted 2012-02-07; First posted 2012-02-09 (Estimated); Last update posted 2012-02-09 (Estimated); Status verified 2012-02

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Time Perspective: Cross-Sectional

GROUPS / COHORTS (2):
- parkinson's disease, young onset
- Normal

SUMMARY:
Parkinson's disease (PD) is the second most frequent neurodegenerative disorder after Alzheimer's disease. It causes motor dysfunctions, such as bradykinesia, resting tremor, rigidity and postural instability. Although PD appears to be sporadic in most cases, several causative genes and susceptibility factors have been identified that cause familial forms of the disease with Mendelian inheritance with autosomal dominant or autosomal recessive inheritance.

Approximately 5~10% of patients with the clinical picture of PD carry a mutation in one of the known genes that cause monogenic forms of the disorder. The average age at onset is between 60 and 80 years and the average age of diagnosis is 60 years. Onset of primary parkinsonism before 50 years is known as early onset parkinsonism(EOP). Onset between 20 and 50 years is known as young-onset PD. Onset at younger than 20 years is known as juvenile parkinsonism (JP). At least, 13 loci and 9 genes are reported. The investigators study is aimed to screen the clinical diagnosed familial EOP for the common mutation site by PCR/DNA sequencing. The gene for screen are Parkin (pattern: PARK2), PINK1 (pattern: PARK6) and ATP13A2 (pattern: PARK9).

ELIGIBILITY:
Inclusion Criteria:

* Idiopathic Parkinson's disease (according to UK Parkinson's Disease Society Brain Bank clinical diagnosis criteria)
* Onset before 50-year-old or positive family history

Exclusion Criteria:

* Secondary parkinsonism

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: patients from China Medical University Hospital
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2012-01

CONTACTS AND LOCATIONS:
Locations (1):
- China Medical University Hospital, Taichung, Taiwan